CLINICAL TRIAL: NCT04533464
Title: MultiStem® for Treatment of Trauma Induced Multiple Organ Failure/Systemic Inflammatory Response Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: Memorial Hermann Hospital (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B06-01
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Trauma; Adult Stem Cells
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MultiStem (Experimental)
  Interventions: Biological: MultiStem
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MultiStem — Intravenous Infusion
  Arms: MultiStem
Biological: Placebo — Intravenous Infusion
  Arms: Placebo

SUMMARY:
Single center, prospective, randomized, double-blind, pragmatic Phase 2 clinical study in severely injured trauma patients within hours of hospitalization who have survived initial resuscitation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older AND
2. Received at least 3 units of any blood product in any hour before Shock Trauma Intensive Care Unit (STICU) arrival AND
3. Survived to initial ICU arrival AND
4. Initial hemostasis has been achieved, in the opinion of the attending surgeon AND
5. Predicted to survive at least 24 hours after STICU arrival by the attending physician AND
6. Ability to start and complete investigational product infusion within 24 hours after known or estimated time of injury.

Exclusion Criteria:

1. Prisoners, defined as those who have been directly admitted from a correctional facility.

   Prisoners are excluded because of their vulnerable population status. A free-living individual who is under police observation as a suspect will remain in the study until discharge or incarcerated.
2. Pregnant and lactating females. It is unknown how stem cells affect a developing fetus or if they can be found in milk. To protect the safety of developing fetuses and breastfeeding children, pregnant and lactating women will be excluded.
3. Have a head injury deemed non-survivable by the trauma or neurosurgery attending. The attending physician may determine futility from a range of injuries/physiological responses. These may include non-survivable TBI (malignant ICP elevation despite maximal therapy with findings of uncal herniation and/or brain dead exam; atlantooccipital dissociation), cardio-pulmonary failure refractory to resuscitation and those patients with an advanced directive that declines resuscitative or organ support therapies.
4. Hemodynamically unstable or requiring clinically meaningful escalation of vasopressor dose for blood pressure support (to maintain SBP ≥ 90 mmHg) during the 30 minute period prior to study product thawing/preparation. Clinically meaningful vasopressor dose adjustment defined as ≥ 5 mcg/min increase in norepinephrine dose; ≥ 50 mcg/min increase in phenylephrine dose; ≥ 5 mcg/kg/min increase in dopamine dose; and ≥ 0.05 mcg/kg/min increase in epinephrine dose. If the patient is on vasopressin, investigators will be instructed not to titrate the vasopressin dose during this 30 minute period.
5. Greater than 20% total body surface area burns and/or suspected inhalation injury.

   Subjects with large and severe thermal injuries and inhalation injures require a resuscitation approach that is different from current isolated trauma resuscitation strategies. Additionally, in the absence of concomitant severe blunt trauma, these subjects are unlikely to receive blood products in the early resuscitative phase.
6. Preexisting chronic kidney disease, defined by prior documented glomerular filtration rate less than 60 mL/min/1.73m2 for 3 months or more. Patients who are unable to communicate their pre-existing conditions will be excluded by Medical Alert bracelets/IDs, stigmata pathognomonic for chronic kidney disease such as presence of dialysis vascular access devices or shunts/markedly elevated BUN/Creatinine, or abdominal incisions consistent with organ transplantation, etc.
7. Preexisting chronic liver disease, evidenced by clinical or laboratory examinations consistent with chronic liver disease/failure (Childs A-C), patient or family report, Medical Alert bracelets/IDs or abdominal incisions consistent with organ transplantation, etc.
8. Known condition of single kidney or concurrent use of potentially nephrotoxic medications at doses likely to be nephrotoxic
9. Known immunodeficient condition or concurrent use of potentially immunosuppressive medications at doses likely to result in an immunosuppressed status
10. Known allergy to MultiStem, dimethyl sulfoxide or human serum albumin
11. No available intravenous access (peripheral or central) of at least 22-guage that can be utilized exclusively for investigational product during the time of planned infusion
12. Clinical condition would be anticipated to deteriorate with intravenous administration of 250 ml of crystalloid
13. Known Do Not Resuscitate (DNR) prior to randomization
14. Enrolled in a concurrent ongoing interventional clinical trial
15. Known functional asplenia or prior surgical removal of the spleen, or a trauma related splenic injury sufficient to precluding enrollment as determined by the PI or Co- Investigators. (trauma related splenic injuries include surgical total splenectomy or nonoperative management of AAST grade V splenic injury including splenic arterial embolization.* *Proximal splenic arterial embolization to control bleeding that leaves the spleen in situ and perfused (below Grade V) does not necessarily exclude the patient. Further, achieving Grade V, with an upgraded score due to a secondary small laceration, etc. away from primary injury will be considered a Grade IV for the purposes of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
A composite of the highest Acute Kidney Injury stage (based on KDIGO guidelines) | Day 30

SECONDARY OUTCOMES:
Mortality | Day 30, Day 90, Day 365
  mortality including median time to death within the acute hospitalization period
Incidence of Acute Kidney Injury adjusted for the competing risk of death | Day 30
Incidence of sepsis, Acute Respiratory Distress Syndrome, Multiple Organ Failure, and Venous Thromboembolism | Day 30
Hospital days | Day 30
  Free days will be defined as the number of days an individual was alive and not in the hospital.
ICU days | Day 30
  Free days will be defined as the number of days an individual was alive and not in the ICU.
ventilator-free days | Day 30
  Free days will be defined as the number of days an individual was alive and not on the ventilator.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cox, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Healios Investigational Site, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No